CLINICAL TRIAL: NCT04160611
Title: Impact of Premedication With Midazolam in Aspiration Procedures On Stress Levels During IVF Procedures
Brief Title: What Amount of Stress is Enough for a Successful Conception?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant Otorhinolaryngologist and Head and Neck Surgeon, University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP-9157/18-14
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: In Vitro Fertilization; Stress; Midazolam Adverse Reaction; Stress, Emotional
Keywords: IVF; stress; midazolam; premedication
MeSH Terms: conditions — Stress, Psychological | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Two randomized groups receiving midazolam/not receiving midazolam premedication before oocyte aspiration procedures as part of IVF procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premedication with Midazolam (Experimental): Patients will be randomly divided into two groups, control and midazolam. The midazolam group will receive midazolam premedication in such a way that 7.5mg midazolam will be taken orally 30 minutes before the aspiration procedure. Because midazolam causes sedation, the woman will be monitored by midazolam after medical premedication to avoid possible complications and will not be allowed to get out of bed on her own for 30 minutes. After 30 min, all women, both test and control group, will begin aspiration under the control of transvaginal ultrasound of one or more mature follicles (TUGOR - transvaginal ultrasound guided oocyte retrieval) under short term general anesthesia.
  Interventions: Drug: Midazolam 7.5mg
- No Premedication with Midazolam (No Intervention): Women in the control group will undergo aspiration under the control of transvaginal ultrasound of one or more mature follicles (TUGOR - transvaginal ultrasound guided oocyte retrieval) under short term general anesthesia.

INTERVENTIONS:
Drug: Midazolam 7.5mg — The patient groups differ only in that respect that the intervention group will receive oral midazolam 7.5 g before oocyte aspiration.
  Arms: Premedication with Midazolam

SUMMARY:
The aim of the study is to determine whether premedication with midazolam before oocyte aspiration in IVF procedures affects the amount of (oxidative) stress in women undergoing IVF and whether stress is also transmitted to the follicular fluid of aspirated follicles. The primary endpoint is the impact of stress during aspiration on the success of medically assisted fertilization (IVF / ICSI in the stimulated cycle).

DETAILED DESCRIPTION:
The procedure of in vitro fertilisation (IVF) is used to treat the infertility problems. The procedure includes ovary aspiration, to isolate oocytes. During the aspiration the patient is sedated with short-term intravenous aesthetic. Premedication is often used in anaesthesiology, and includes drugs application 30 minutes prior to procedure to sedate and treat the anxieties of the patient. One of the most often used drugs in premedication is midazolam. As the procedure is quite stressful for the patients, our aim is to investigate the influence of midazolam premedication on the stress release during the oocyte aspiration procedure, as well as its influence on the whole IVF procedure. Therefore, patients will be divided into two groups, control and midazolam. Blood samples will be taken before and during the procedure. Stress, antioxidant parameters (with glutathione and catalase) and oxidative status will be monitored in serum and follicular fluid.

The results will be correlated with subjective stress levels in the two groups in an effort to establish ties with IVF results.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, healthy women undergoing IVF procedures for the first time

Exclusion Criteria:

* Refusal to enroll, chronic endocrine and psychiatric illnesses that might affect baseline stress levels

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female - IVF procedure related
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Stress Levels in Premedicated Women | 3 hours post-surgery
  All patients in the midazolam group will be sampled with 5 ml venepuncture prior to midazolam administration, just before the procedure, 2 hours after the procedure. A follicular fluid sample will be taken at the procedure. Samples will be stored in the freezer at -80⁰C. The total antioxidant capacity (TAC) and total oxidation capacity (TOC) of commercially available kits will be determined from plasma and follicular fluid. Whole blood will determine total glutathione and catalase activity. In addition to the total oxidation capacity, the amount of HNE-protein conjugates will be determined from the follicular fluid as an indicator of lipid peroxidation, and the Patients will be monitored after the aspiration procedure, and the success of the procedure of medically assisted fertilization, ie number of pregnancies, in the test and control group will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Košec, MD, PhD, Study Chair — Department of Gynecology and Obstetrics, University Hospital Center Sestre milosrdnice, Zagreb, Croatia
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No